CLINICAL TRIAL: NCT04388540
Title: Caribbean Island Urinary Iodine Survey 2018
Acronym: CRUISE
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Pan American Health Organization (Other); UNICEF (Other)
Responsible Party: Sponsor
Other Study IDs: CRUISE
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Iodine Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Spot Urine Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Jamaica: School aged children 6 - 12 years living in Jamaica
- Trinidad and Tobago: School aged children 6 - 12 years living in Trinidad and Tobago
- Belize: School aged children 6 - 12 years living in Belize
- Barbados: School aged children 6 - 12 years living in Barbados
- St. Lucia: School aged children 6 - 12 years living in St. Lucia
- Grenada: School aged children 6 - 12 years living in Grenada
- St. Vincent & the Grenadines: School aged children 6 - 12 years living in St. Vincent & the Grenadines
- Antigua: School aged children 6 - 12 years living in Antigua
- Dominica: School aged children 6 - 12 years living in Dominica
- St. Kitts and Nevis: School aged children 6 - 12 years living in St. Kitts and Nevis

SUMMARY:
Many of the Caribbean island nations have no data on iodine status in their populations.

Iodine deficiency in children can reduce IQ but can be easily corrected through a program of salt iodization.

The study will be located at 11 islands of the Caribbean region. At each of the 11 study sites, we will measure the iodine status in school-age children by collecting morning spot urine samples for measurement of urinary iodine concentration (UIC). We will also measure height and weight in all children. We will collect a repeat, next-day spot urine sample in 1/3rd of children to adjust for intra-individual variation in spot UIC and calculate the distribution of population intake.

DETAILED DESCRIPTION:
In well-controlled randomized trials in Europe and New Zealand, even mild-to-moderate iodine deficiency in school-age children reduces IQ (1); thus, its critical to avoid iodine deficiency in this age group. In countries effected by iodine deficiency, its sustainable elimination through iodized salt can contribute to socioeconomic development. The goal to eliminate iodine deficiency was first adopted globally at the World Summit for Children in 1990, and in 1994, WHO and UNICEF concluded that salt iodization is a safe, cost-effective and sustainable strategy to control iodine deficiency (2). In 2005, the World Health Assembly called on national governments to report on their iodine nutrition every three years. However, before the present survey, the ten countries included in this project had no data on iodine status in their populations, and household access to adequately iodized salt was also unknown. Thus, the study objectives were:

* Assess the distribution of iodine intake of school-age children and their iodine status by measuring urinary iodine concentrations;
* Assess the iodine content of household salt and of seasoning powders;
* Based on the above, provide the preliminary evidence base on which to make initial recommendations for iodine strategy/programs in the region.

ELIGIBILITY:
Inclusion Criteria:

1. age at study enrolment 6 to 12 years
2. healthy; no known history of major medical illnesses and taking no chronic medications;
3. residence at the respective study site for 12 months or longer;
4. no use of iodine containing dietary supplements during the last 6 months;
5. no use of X-ray / CT contrast agent or iodine containing medication within the last year.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children of school age
Sampling Method: Non-Probability Sample
Enrollment: 3080 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Iodine status (UIC in spot urine samples) | March 2018 to May 2019
  Assessment of iodine status based on median urinary iodine concentration in spot urine samples

SECONDARY OUTCOMES:
Iodine content in salt | January 2019 to May 2019
  Measurement of iodine concentration in salt samples brought in by participants

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Dr. Prof., Principal Investigator — ETH Zurich, Iodine Global Network
Locations (10):
- Pan American Health Organization, St John's, Antigua and Barbuda
- Pan American Health Organization, Bridgetown, Barbados
- Ministry of Health, Belize City, Belize
- Pan American Health Organization, Roseau, Dominica
- Pan American Helath Organization, The Lime, Grenada
- The University of the West Indies, Mona, Kingston, Jamaica
- Ministry of Health, Basseterre, Saint Kitts and Nevis
- Ministry of Health and Wellness, Castries, Saint Lucia
- Pan American Health Organization, Kingstown, Saint Vincent and the Grenadines
- University of the West Indies, Port of Spain, Trinidad and Tobago